CLINICAL TRIAL: NCT02430233
Title: Vaginal Progesterone for the Prolongation of Pregnancy After Arrested Pre-term Labor - Randomized Double Blind Placebo Controlled Trial
Brief Title: Vaginal Progesterone for the Prolongation of Pregnancy After Arrested Pre-term Labor
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: HaEmek Medical Center, Israel (Other)
Responsible Party: Principal Investigator, Zohar Nachum, Principal Investigator, HaEmek Medical Center, Israel
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0080-13
Record Dates: First submitted 2015-04-20; First posted 2015-04-30 (Estimated); Last update posted 2023-02-28 (Actual); Status verified 2023-02

CONDITIONS: Preterm Labor
MeSH Terms: conditions — Obstetric Labor, Premature | interventions — Progesterone; Utrogestan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- micronized progesterone 400 mg (Experimental): participants receive vaginal micronized progesterone (Utrogestan- 200mg×2 PV(per vagina) per day)
  Interventions: Drug: micronized progesterone 400 mg (Utrogestan)
- No treatment (No Intervention): No treatment

INTERVENTIONS:
Drug: micronized progesterone 400 mg (Utrogestan) — participants receive vaginal micronized progesterone (Utrogestan- 200mg×2 PV(per vagina) per day)
  Other Names: Utrogestan- 200mg×2 PV(per vagina) per day
  Arms: micronized progesterone 400 mg

SUMMARY:
Patients diagnosed with arrested pre-term labor following tocolytics at 24-34 gestational weeks will be randomly allocated to receive either vaginal micronized progesterone 400 mg/day or no treatment.

DETAILED DESCRIPTION:
Since progesterone derivatives are useful in preventing preterm labor in cases of risk factors or previous preterm labor, we hypothesize that they will also show efficacy in pregnancy prolongation in women whose preterm labor was arrested following tocolytic treatment.

Patients diagnosed with arrested pre-term labor following tocolytics at 24-34 gestational weeks will be randomly allocated to receive either vaginal micronized progesterone 400 mg/day or no treatment.

This study has the potential to find a treatment to prevent preterm labor and thus to reduce neonatal morbidity and mortality.

ELIGIBILITY:
Inclusion Criteria:

1. 18 years of age
2. Tocolytic treatment between 24+0 and 34+0 weeks
3. Patient's consent to participate in this study
4. 24 hours after tocolytic initiation and up to 3 days after finishing the tocolytic treatment
5. Arrest of preterm labor

Exclusion Criteria

1. Contraindication to ongoing pregnancy including:

   1. Suspected amnionitis during testing for eligibility- evidence of active infection including temperature ≥ 38.0°C and uterine tenderness, foul-smelling vaginal discharge, maternal tachycardia of 120 beats per minute or greater, or sustained fetal tachycardia of 160 beats per minute or greater
   2. Evidence of significant placental abruption (contractions and significant bleeding from placental origin)
   3. Intrauterine fetal death diagnosed at the time of admission
2. Major fetal malformation
3. Known maternal allergy to progesterone
4. Current use of progesterone at the time of admission
5. Epilepsy
6. Breast cancer
7. PPROM (preterm premature rupture of membranes) during testing for eligibility
8. Age below 18 years
9. Known active liver disease (elevated liver enzymes at twice the upper normal limit according to medical history or blood test that were taking doring standard medical care)
10. History of deep vein thrombosis
11. Major active psychiatric disorders (major affective disorders and psychotic disorders)
12. Uncontrolled chronic hypertension
13. Heart failure
14. Chronic renal failure
15. Pre-gestational diabetes with known target organ damage
16. History of spontaneous preterm delivery
17. Previous tocolytic treatment during the current pregnancy

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 129 (Actual)
Dates: Start 2018-12-19 (Actual); Primary Completion 2023-02-27 (Actual); Study Completion 2023-02-27 (Actual)

PRIMARY OUTCOMES:
The mean number of days from enrollment to delivery | Up to 18 weeks
The rate of preterm spontaneous delivery | Up to 13 weeks
  defined as spontaneous labor or preterm delivery following induction/cesarean section due to preterm premature rupture of membranes prior to 37 weeks of gestation

SECONDARY OUTCOMES:
Number of days from recruitment to repeated preterm labor episode or preterm premature rupture of membranes, up to 37 weeks of gestation | Up to 13 weeks
Pregnancy prolongation beyond one week | Up to 18 weeks
Need for repeated acute tocolysis | Up to 13 weeks
Number of hospitalizations and length of stay until 36.6 gestational weeks | Up to 13 weeks
The rate of preterm spontaneous labor (defined as spontaneous labor or preterm premature rupture of membranes prior to 37 weeks of gestation) | Up to 13 weeks
Admission to the NICU (neonatal intensive care unit) | From delivery and up to 28 days
Length of NICU stay | From delivery and up to 3 months
Length of neonate hospital stay | From delivery and up to 3 months
Fetal/neonatal death | Around delivery
Birth weight and the rate of small for gestational age neonates | Around delivery
The rate of neonatal complications | From delivery and up to 3 months
  including transient tachypnea, RDS (respiratory distress syndrome), bronchopulmonary dysplasia, ventilatory support, supplemental oxygen, IVH (intraventricular hemorrhage), NEC (necrotizing enterocolitis), PDA (patent ductus arteriosus), retinopathy, neonatal sepsis, and congenital abnormalities not previously identified (specifically genital abnormalities).
The rate of chorioamnionitis and endometritis | around delivery and up to 1 week post-partum
Adverse medication reactions | Up to 13 weeks
Postpartum hemorrhage | From delivery and up to 1 week post-partum
Revision of uterine and cervix and reasons for the procedure | During the 48 hours from delivery
Urinary tract or vulvovaginal infection until 36.6 weeks | Up to 13 weeks

CONTACTS AND LOCATIONS:
Locations (3):
- Israel (3):
  - Poriya Medical Center, Tiberias, North
  - Emek Medical center, Afula, Please Select
  - Assuta Ashdod medical center, Ashdod

REFERENCES:
- [Derived] Nachum Z, Ganor Paz Y, Massalha M, Wated M, Harel N, Yefet E. Vaginal Progesterone for Pregnancy Prolongation After Arrested Preterm Labor: A Randomized Clinical Trial. JAMA Netw Open. 2024 Jul 1;7(7):e2419894. doi: 10.1001/jamanetworkopen.2024.19894. PMID 38976270